CLINICAL TRIAL: NCT01374971
Title: Open-Label Pre and Post Treatment Arthroscopic Synovial Biopsy Study for the Assessment of Certolizumab Pegol Immunomodulatory Synovial Effects on Select Biomarkers and Gene Expression
Brief Title: Rheumatoid Arthritis Treatment and Biopsy Study Assessing Certolizumab Pegol (Cimzia)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nathan Wei, MD, FACP, FACR: (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor-Investigator, Nathan Wei, MD, FACP, FACR:, Nathan Wei, MD, FACP, FACR, Arthritis Treatment Center, Maryland
Organization: Arthritis Treatment Center, Maryland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ATC2011
Record Dates: First submitted 2011-06-14; First posted 2011-06-17 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Cimzia; Certolizumab Pegol; Arthroscopic Synovial biopsy; Office Based Procedure; Biologic; Tumor Necrosis Factor (TNF); Anti-TNF
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Certolizumab Pegol (CZP) (Other): Certolizumab Pegol (CZP) liquid formulation 200 mg sc -(initial loading dose of 400 mg sc at 0 (Baseline), 2, and 4 weeks), then 200 mg sc every 2 weeks at 6, 8, and 10 weeks with arthroscopic synovial tissue biopsy pre- and post-treatment.
  Interventions: Drug: Certolizumab Pegol (CZP); Procedure: Arthroscopic synovial tissue biopsy

INTERVENTIONS:
Drug: Certolizumab Pegol (CZP) — CZP is an anti-TNF, humanized antibody Fab' fragment/polyethylene glycol(PEG)conjugate. CZP liquid formulation 200 mg sc -(initial loading dose of 400 mg sc at 0 (Baseline), 2, and 4 weeks), then 200 mg sc every 2 weeks at 6, 8, and 10 weeks.
  Other Names: Brand Name: Cimzia; UCB product: Certolizumab Pegol (CDP870); Pre-filled syringe: NDC50474-710-79
Procedure: Arthroscopic synovial tissue biopsy — Subjects will undergo arthroscopy Pre and Post Treatment. The arthroscopy will be performed on a clinically inflamed joint. A single arthroscopy procedure using a small bore arthroscope will be conducted to obtain synovial tissue in each joint in all subjects. Local anesthesia will be used only. Two small incisions will be made to accommodate the arthroscope and other instruments. Synovial biopsies will be obtained using a motorized shaver.

SUMMARY:
The purpose of this study is to conduct an Investigator-Sponsored Study to determine the potential immunomodulatory effects of Certolizumab Pegol (CZP) treatment at the site of disease activity (synovial lining) in subjects with rheumatoid arthritis (RA), using pre treatment and post treatment arthroscopic synovial biopsies and ex vivo on gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent document
* Subjects must be at least 18 years of age or older
* Subject must be willing and able to comply with scheduled visits, arthroscopy, laboratory tests, and other procedures
* Diagnosis of RA based on American College of Rheumatology (ACR) 1987 Revised Criteria
* Active disease at screening visit
* Methotrexate taken continuously for at least 12 weeks at a stable dosage
* Sexually active women of child-bearing potential and men whose partners are women of child-bearing potential are required to use adequate contraceptive methods during participation on this trial
* Treatment with non-steroidal anti-inflammatory drugs (NSAIDS)and oral corticosteroids (less than or equal to 10 mg/day prednisone or equivalent)is accepted

Exclusion Criteria:

* Diagnosis of any other inflammatory arthritis
* History of infected joint prosthesis that is still in situ
* History of allergy to local anesthetic agents
* Pregnant or lactating women
* Current or recent history of uncontrolled clinically significant conditions(e.g..,kidney disease, liver disease, class III or IV congestive heart failure, according to the New York Heart Association)
* History or suspected demyelinating disease of the central nervous system, e.g. multiple sclerosis or optic neuritis
* Current participation in clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Wei, MD,FACP,FACR, Principal Investigator — Nathan Wei, MD, PA d/b/a Arthritis Treatment Center, 301-694-5800
Locations (1):
- Arthritis Treatment Center, Frederick, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Certolizumab Pegol (CZP): Certolizumab Pegol (CZP) liquid formulation 200 mg sc -(initial loading dose of 400 mg sc at 0 (Baseline), 2, and 4 weeks), then 200 mg sc every 2 weeks at 6, 8, and 10 weeks.
  Certolizumab Pegol (CZP): CZP is an anti-Tumor Necrosis Factor (TNF), humanized antibody Fab' fragment/polyethylene glycol(PEG)conjugate. CZP liquid formulation 200 mg sc -(initial loading dose of 400 mg sc at 0 (Baseline), 2, and 4 weeks), then 200 mg sc every 2 weeks at 6, 8, and 10 weeks.
  Arthroscopic synovial tissue biopsy: Subjects will undergo arthroscopy Pre and Post Treatment. The arthroscopy will be performed on a clinically inflamed joint. A single arthroscopy procedure using a small bore arthroscope will be conducted to obtain synovial tissue in each joint in all subjects. Local anesthesia will be used only. Two small incisions will be made to accommodate the arthroscope and other instruments. Synovial biopsies will be obtained using a motorized shaver.
Period: Overall Study
Arm/Group | Certolizumab Pegol (CZP)
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All subjects who meet screening criteria were enrolled until target number of 12 subjects was met.
Groups:
- Certolizumab Pegol (CZP): Certolizumab Pegol (CZP) liquid formulation 200 mg sc -(initial loading dose of 400 mg sc at 0 (Baseline), 2, and 4 weeks), then 200 mg sc every 2 weeks at 6, 8, and 10 weeks.
  Certolizumab Pegol (CZP): CZP is an anti-TNF, humanized antibody Fab' fragment/polyethylene glycol(PEG)conjugate. CZP liquid formulation 200 mg sc -(initial loading dose of 400 mg sc at 0 (Baseline), 2, and 4 weeks), then 200 mg sc every 2 weeks at 6, 8, and 10 weeks.
  Arthroscopic synovial tissue biopsy: Subjects will undergo arthroscopy Pre and Post Treatment. The arthroscopy will be performed on a clinically inflamed joint. A single arthroscopy procedure using a small bore arthroscope will be conducted to obtain synovial tissue in each joint in all subjects. Local anesthesia will be used only. Two small incisions will be made to accommodate the arthroscope and other instruments. Synovial biopsies will be obtained using a motorized shaver.
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 12
Age, Customized [Number; unit: years]
  >18 years of age | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Synovial TNFa, CXCL13, IL-8, IL-6, IL-1b, IL-10, IP-10, BCL3, CD3E, DUSP4, FOXP3, CD79A, CD138, MMP-3, and MMP-1 After 12 Weeks of Treatment With Certolizumab Pegol (CZP) in Patients With Rheumatoid Arthritis
Description: Synovial tissue biopsy samples were taken at baseline and at 12 weeks after starting treatment with CZP. These samples were analyzed to determine the concentrations of select biomarkers and to determine the percent change in concentration from baseline to week 12.
Time Frame: Baseline and Week 12
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 11
Percent change
  TNFa | -10.1 [-23.4 to 3.2]
  CXCL13 | -53.4 [-69.0 to -37.8]
  IL-8 | 128.5 [22.9 to 234.1]
  IL-6 | -3.3 [-27.8 to 21.2]
  IL-1b | 91.7 [10.1 to 173.3]
  IL-10 | 204.8 [48.3 to 361.3]
  IP-10 | 8.7 [-37.6 to 55.0]
  BCL3 | -32.4 [-38.5 to -26.3]
  CD3E | -17.5 [-37.8 to 2.8]
  DUSP4 | -13.5 [-33.4 to 6.4]
  FOXP3 | -2.3 [-27.4 to 22.8]
  CD79A | 110.4 [31.9 to 188.9]
  CD138 | 111.9 [52.5 to 171.3]
  MMP-3 | -44.9 [-57.9 to -31.9]
  MMP-1 | -67.9 [-76.5 to -59.3]

2. Secondary Outcome: Percent Change From Screening in Disease Activity Score (DAS) 28 ESR After 14 Weeks of Treatment
Description: The DAS 28 ESR is a score calculated from the results of a 28-count joint assessment (total number of tender joint possible is 28, and total number of swollen joints possible is 28), the Erythrocyte Sedimentation Rate (ESR), and the Patient Global Assessment (measured using a 100 mm visual analogue scale, with the lowest possible score of 0 mm meaning the subject is not affected at all by arthritis and the highest possible score of 100 mm meaning the subject is severely affected by arthritis). A lower DAS 28 ESR indicates less active disease, and a higher DAS 28 ESR indicates more active disease. The DAS 28 ESR was calculated for each subject at the screening visit and at the Week 14 final visit. The percent change was then calculated for each patient, and a mean percent change for all subjects was determined.
Time Frame: Screening and Week 14
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 12
percent change | -27.5 (25.3)

ADVERSE EVENTS:
Arm/Group | Certolizumab Pegol (CZP)
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (CZP) (N=12)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Flare of Rheumatoid Arthritis (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes